CLINICAL TRIAL: NCT00765856
Title: An Open-Label Safety and Tolerability Study of Immediate-Release and Extended-Release Oxymorphone in Opioid-Tolerant Pediatric Subjects With Chronic Pain.
Brief Title: Open-Label Safety and Tolerability of Oxymorphone IR and ER in Opioid Tolerant Pediatric Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated new protocol developed which incorporated Pharmacokinetics
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3202 036
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
Keywords: Opioid tolerant; Pediatric; Male 6-17 years of age; Female 6-17 years of age; Pain; Non malignant; Malignant
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxymorphone ER (Experimental)
  Interventions: Drug: Oxymorphone ER

INTERVENTIONS:
Drug: Oxymorphone ER — Oxymorphone ER dosing adjustments made under the direction of the Investigator during the Titration Period.
  Oxymorphone IR (Opana) IR 5mg tablet - used as rescue medications
  Other Names: Opana ER, Opana

SUMMARY:
Patients will convert from current opioid to Oxymorphone ER and undergo titration. During the Titration Period, subjects will receive daily oxymorphone Extended Release tablets(s) every 12 hours. Dosing adjustments will be based on the review of the subject's pain scores. Oxymorphone IR 5 mg will be provided to be used as supplemental "breakthrough" pain medication (as needed). Titration Period will end when the fixed dose of study medication is tolerated and the subject achieves adequate analgesia. Subjects will then proceed to the open-label 3-month maintenance period on the fixed dose of study medication established during the Titration Period.

DETAILED DESCRIPTION:
An Open-Label Safety and Tolerability Study of Immediate-Release and Extended-Release Oxymorphone in Opioid-Tolerant Pediatric Subjects With Chronic Pain.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic cancer or non-cancer pain, currently requiring treatment of pain with a strong opioid for at least 5 days (3 of 5 days at a dose greater than or equal to 45 mg/daily (qd) oral morphine equivalent)
* Weigh at least 50 kg
* Expected to continue to require a strong opioid for pain relief for at least 4 weeks and up to 4 months.

Exclusion Criteria:

* Have a life expectancy <4 weeks
* Plan to undergo a surgical procedure within 3 days of study entry or during the Titration Period
* Have dysphagia or difficulty swallowing whole tablets
* Have a previous exposure to oxymorphone
* Have an ileostomy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2010-02-22 (Actual); Study Completion 2010-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director CR&D, Study Director — Endo Pharmaceuticals
Locations (13):
- United States (13):
  - Arkansas Childrens's Hospital-Division of Pediatric Anestesia and Pain Medicine, Little Rock, Arkansas
  - Stanford University School of Medicine, Stanford, California
  - The Children's Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Tukoi Clinical Research, Miami, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Taylor Research, LLC, Marietta, Georgia
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - University of Louisville Reserach Foundation, Inc., Louisville, Kentucky
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Hershey Medical Center, Hershey, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymorphone ER: Oxymorphone ER dosage was adjusted by investigator during the titration period. Study was terminated early by the Sponsor.
Period: Titration Period
Arm/Group | Oxymorphone ER
Started | 27
Completed | 24
Not Completed | 3
Period: Maintenance Period
Arm/Group | Oxymorphone ER
Started | 24
Completed | 18
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Oxymorphone ER: Open-label dose titration period of up to 4 weeks and open-label maintenance period of up to 12 weeks.
Arm/Group | Oxymorphone ER
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 2
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Extent of Exposure to Oxymorphone Extended-Release: Average Daily Dose
Description: Data based on drug accountability data from the case report forms. Data is based on the number of enrolled participants in each treatment period. All participants entering maintenance period finished titration period. Study was terminated early by Sponsor due to a change in the FDA postmarketing requirement. The study was not terminated for safety reasons.
Time Frame: Day 1 up to Day 112 (approximately 4 weeks for titration period and 12 weeks for the maintenance period)
Population: Safety population defined as all participants that took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Titration Period: Open-label dose titration period of up to 4 weeks
- Maintenance Period: Open-label maintenance period of up to 12 weeks
Arm/Group | Titration Period | Maintenance Period
Number analyzed (Participants) | 27 | 24
mg | 35.25 (11.955) | 39.11 (15.176)

2. Secondary Outcome: Extent of Exposure to Oxymorphone Extended-Release: Total Number of Tablets Taken
Description: as for outcome 1
Time Frame: Day 1 up to Day 112 (approximately 4 weeks for titration period and 12 weeks for the maintenance period)
Population: Safety population defined as all participants that took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Titration Period | Maintenance Period
Number analyzed (Participants) | 27 | 24
Tablets | 36.1 (15.63) | 162.7 (66.77)

3. Secondary Outcome: Extent of Exposure to Oxymorphone Immediate-Release Rescue Medication: Total Daily Dose
Description: Data based on drug accountability data from the case report forms. Data with missing dates are included in calculation. Data is based on the number of enrolled participants in each treatment period. Two (2) participants did not use Oxymorphone IR as rescue medication in the Titration period. Therefore, 25 out of 27 participants were analyzed for this outcome measure. All participants entering maintenance period finished titration period. Study was terminated early by Sponsor due to a change in the FDA postmarketing requirement. The study was not terminated for safety reasons.
Time Frame: Day 1 up to Day 112 (approximately 4 weeks for titration period and 12 weeks for the maintenance period)
Population: Safety population defined as all participants that took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Titration Period: Open-label dose titration period of up to 4 weeks. Two (2) participants did not use Oxymorphone IR as rescue medication in the Titration period. Therefore, 25 out of 27 participants were analyzed for this outcome measure
Arm/Group | Titration Period | Maintenance Period
Number analyzed (Participants) | 25 | 24
mg | 7.9 (3.01) | 5.5 (1.49)

4. Secondary Outcome: Extent of Exposure to Oxymorphone Immediate-Release Rescue Medication: Average Number of Daily Rescues
Description: Average number of daily rescues per day by participants. Data based on drug accountability data from the case report forms. Data with missing dates are included in calculation. Data is based on the number of enrolled participants in each treatment period. Two (2) participants did not use Oxymorphone IR as rescue medication in the Titration period. Therefore, 25 out of 27 participants were analyzed for this outcome measure. All participants entering maintenance period finished titration period. Study was terminated early by Sponsor due to a change in the FDA postmarketing requirement. The study was not terminated for safety reasons.
Time Frame: Day 1 up to Day 112 (approximately 4 weeks for titration period and 12 weeks for the maintenance period)
Population: Safety population defined as all participants that took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Rescue doses/day
Arm/Group | Titration Period | Maintenance Period
Number analyzed (Participants) | 25 | 24
Rescue doses/day | 1.5 (0.45) | 1.1 (0.30)

5. Secondary Outcome: Extent of Exposure to Oxymorphone Immediate-Release Rescue Medication: Total Number of Doses
Description: Total number of doses (Tablets) taken by participants. Data based on drug accountability data from the case report forms. Data with missing dates are included in calculation. Data is based on the number of enrolled participants in each treatment period. Two (2) participants did not use Oxymorphone IR as rescue medication in the Titration period. Therefore, 25 out of 27 participants were analyzed for this outcome measure. All participants entering maintenance period finished titration period. Study was terminated early by Sponsor due to a change in the FDA postmarketing requirement. The study was not terminated for safety reasons.
Time Frame: Day 1 up to Day 112 (approximately 4 weeks for titration period and 12 weeks for the maintenance period)
Population: Safety population defined as all participants that took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Total number of doses
Arm/Group | Titration Period | Maintenance Period
Number analyzed (Participants) | 25 | 24
Total number of doses | 19.0 (15.36) | 17.4 (40.60)

ADVERSE EVENTS:
Time Frame: First dosing up to 30 days after the last dose of study medication, approximately 20 weeks (titration period of up to 4 weeks, the maintenance period of up to 12 weeks and 30 days post-last dose).
Groups:
- Maintenance Period: Open-label maintenance period of up to 12 weeks plus 30 days post-last dose
Arm/Group | Titration Period | Maintenance Period
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/27 | 3/24
Other Adverse Events (participants affected / at risk) | 15/27 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Titration Period (N=27) | Maintenance Period (N=24)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 0 | 1
Acute pancreatitis (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased alanine aminotransferase (Investigations) | 0 | 1
Increased aspartate aminotransferase (Investigations) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Pouchitis (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Titration Period (N=27) | Maintenance Period (N=24)
Somnolence (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No